CLINICAL TRIAL: NCT05322291
Title: The Effect of Mobile-Based Training and Counseling Developed for Hemodialysis Patients on Adaptation to the Experienced Symptoms and Disease
Brief Title: The Effect of the Mobile Application Developed for Hemodialysis Patients on Symptoms and Disease Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge AKBABA (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Ozge AKBABA, PhD Student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OAKBABA
Record Dates: First submitted 2022-01-31; First posted 2022-04-11 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Chronic Kidney Failure
Keywords: hemodialysis; Treatment Compliance; symptom managemen; mobile application; chronic kidney failure
MeSH Terms: conditions — Kidney Failure, Chronic; Patient Compliance

STUDY DESIGN:
Intervention Model Description: The mobile application developed will be installed on the phones of hemodialysis patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The developed mobile application will be installed on the phones of hemodialysis patients in the experimental group. Online consultancy and training will be provided with the application.
  Interventions: Behavioral: Mobil Application
- Control Group (No Intervention): No intervention will be made. They will continue to receive routine care.

INTERVENTIONS:
Behavioral: Mobil Application — The mobile application developed will be installed on the phones of hemodialysis patients
  Arms: Experimental Group

SUMMARY:
The aim of this study is to determine the effect of mobile-based education and counseling developed for hemodialysis patients on the symptoms experienced and the adaptation to the disease.

DETAILED DESCRIPTION:
Patients with end-stage renal disease are faced with many symptoms both during the disease and during the hemodialysis treatment process. Likewise, this process brings with it problems of adaptation to the disease. Experiencing intense symptoms negatively affects compliance with the disease and hemodialysis treatment, and compliance problems complicate symptom management. Therefore, patients need information support that can increase symptom management and compliance. Considering today's technology, this information can be provided by mobile phone, especially due to ease of use and fast transportation. In order for patients to access accurate information and receive consultancy from experts, appropriate software and sustainable mobile applications must be included in the disease management process. Today, mobile applications are an integral part of daily life for millions of users worldwide and are increasingly used to receive and communicate fast and interactive information about various chronic diseases. With the mobile-based training and counseling to be applied in this study, it is aimed to enable patients receiving hemodialysis treatment to access professional information support more easily, to better manage the symptoms they experience due to the disease, and to increase their adaptation to the disease. For this reason, the effect of mobile-based training and counseling developed for patients receiving hemodialysis treatment on the symptoms experienced by the patients and their adaptation to the disease will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney failure patient
* Agreeing to be a voluntary participant,
* Receiving dialysis treatment for at least 3 months,
* 18 years and over,
* Able to understand and speak Turkish
* At least primary school graduate,
* Using a smart phone for at least one year,
* Having internet access at home or at work.
* Able to use internet

Exclusion Criteria:

* Speech, hearing and visual impairment,
* Having any psychiatric diagnosis or treatment that may interfere with perception (Alzheimer, schizophrenia, major depression)
* rheumatological diseases, fracture, joint health problem, amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Measure | 0-3 months
  The effect of mobile-based application and counseling on symptom management will be measured in patients receiving hemodialysis treatment. Patient Information Form and Dialysis Symptom Index will be used for measurement. The dialysis symptom scale includes 30 symptoms that describe physical or emotional symptoms. The patient responds to the symptoms he has experienced in the last week as yes-no, no, he/she answers that he/she has not experienced the symptom, and if yes, he/she has the symptom. If your answer is yes, the extent to which this symptom affects the patient is evaluated with a five-point Likert type scale. It is evaluated and scored as 1=none, 5=very much. After the obtained scores are summed, the total scale score is obtained. The scale point ranges from 0-150. The fact that the total score approaches 150 indicates that the effect of the symptom has increased.
Dialysis symptom | 0-3 months
  Reducing dialysis symptoms.

SECONDARY OUTCOMES:
Measure | 3-6 months
  The effect of mobile-based application and counseling on treatment compliance will be measured in patients receiving hemodialysis treatment. Patient Information Form and End Stage Renal Failure Compliance Scale will be used.This 6-item scale, which questions participation in hemodialysis, drug use, fluid restriction and adherence to diet, constitutes the compliance behaviors sub-dimension. The weight system used in scoring these items was determined according to the degree of importance related to the clinical outcome of each section. Items 14, 17, 18, 26, 31 and 46, which evaluate the patient's compliance behaviors, and 15, 19 and 27, which affect the scoring of three of these items, were used in the scale. The total score that can be obtained from the scale is between 0 and 1200. The higher the score, the higher the level of adherence to treatment.
End Stage Renal Failure Compliance | 3-6 months
  End Stage Kidney Failure Improving compliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yıldırım University, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No